CLINICAL TRIAL: NCT05744323
Title: Effects of Functional Training on Fundamental Motor Skills Among Chinese Children Aged 6-7 Years Old in Tai Yuan
Brief Title: Effects of Functional Training on Fundamental Motor Skills Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Dong (Other)
Responsible Party: Sponsor-Investigator, Zhang Dong, Principal Investigator, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CN20230101
Record Dates: First submitted 2023-02-09; First posted 2023-02-27 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Healthy Children
Keywords: functional training

STUDY DESIGN:
Intervention Model Description: The study will be conducted using a randomized controlled trial (RCT), and the study will be divided into three parts: pre-study baseline testing, intervention training and post-study testing. The entire experiment will be conducted in the first academic year of 2023.2-2023.4. A pilot study will be carried out first, followed by the actual research, in order to provide the framework and offer support for the full-scale experiment that will follow. The subjects involved in this study are 6-year-old and 7-year-old children, all students participating in the study will be divided into experimental and control groups.
Who Masked: Participant
Masking Description: in order to avoid the Contamination caused by the mutual interference between the experimental group and the control group, blinding was necessary in the study. In this study, a single-blind experiment will be used to blind the participating children. During sample selection and grouping, the participating children will not know the specific grouping situation, and will not be informed of the relevant experimental objectives
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will engage in functional training
  Interventions: Other: Functional training
- Control group (No Intervention): the control group will follow the state-mandated physical education curriculum.

INTERVENTIONS:
Other: Functional training — Physical and motor function training for children,may use BOSU balls, medicine balls, balance mats, fitness steps, and other training equipment to improve gradually
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to examine the effects that functional training may have on the development of fundamental motor skills and to create a systematic functional training program suitable for healthy children aged 6-7 years.

The main question[s] it aims to answer are:

* [To examine the effects of functional training on FMS among children aged 6-7 years.]
* [To compare the effects of functional training on FMS between boys and girls]

This study will include an experimental group and a control group. The experimental group will engage in functional training, while the control group will follow the state-mandated physical education curriculum. Through experiments, we will investigate the effect of functional training on children's fundamental motor skills and assess whether the experimental group's intervention effect is superior to the control group. The samples in this study were normal Chinese children aged 6-7 years. There were 40 people in both the experimental and control groups, including 20 boys and 20 girls

DETAILED DESCRIPTION:
Training intervention information This study will include an experimental group and a control group. The experimental group will engage in functional training, while the control group will follow the state-mandated physical education curriculum. Through experiments, we will investigate the effect of functional training on children's fundamental motor skills and assess whether the experimental group's intervention effect is superior to the control group. The samples in this study were normal Chinese children aged 6-7 years. There were 66 people in both the experimental group and control groups, including 35 boys and 35 girls.

Training Intervention Protocol for experiment group The selection of training items and content and the design of the training plan are based on the training content and principals involved in books such as the physical and motor function training for children, edited by Zhang Xiuli et al. (2018), the physical function training manual for adolescents and children edited by Wang Xiong (2019), and the functional training edited by Santana (2016). Furthermore, based on the literature review, the training frequency for the experiment was two (2) times a week, each lasting 45 minutes, including a 5-minute warm-up phase, a 35-minute main training phase, and a 5-minute relaxation phase, for a total training time of 12 weeks. The content was changed every two (2) weeks, and the intensity of the main phase of training ranged from 60% to 70%.

Training Intervention Protocol for control group The training content of the control group will be selected by the Compulsory Education Physical Education and Health Curriculum Standard in the year 2022. This standard follows the school's physical education teaching plan; the students in the control group will participate in the school's standard physical education curriculum. The specific content will be based on the actual physical education curriculum of the school. The training frequency for the control group was two times (2) a week, each lasting 45 minutes, and for a total training time of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese Children in Taiyuan
2. Primary school children are aged 6-7
3. Including both gender boys and girls

Exclusion Criteria:

1. Children cannot normally participate in regular physical education courses.
2. The children have movement disorders.
3. The children have physical or mental diseases.
4. During the training period, the children have to do other sports training.

The procedure for selecting samples will make use of stratified sampling in addition to a random number table.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Use the TGMD-2 scale to test locomotor skills | baseline, pre-intervention/Change from baseline locomotor skills at 12 weeks.
  6 patterns tested within locomotor subtests. The scoring is based on points listed for each pattern. The total score is 24 points. The athletic performance will be criterion-based scores compared with norm-referenced standards.
Use the TGMD-2 scale to test object control skills | baseline, pre-intervention/Change from baseline object control skills at 12 weeks.
  6 patterns tested within object control subtests. The scoring is based on points listed for each pattern. The total score is 24 points. The athletic performance will be criterion-based scores compared with norm-referenced standards.
Use the Y-test to test balance skill | baseline, pre-intervention/Change from baseline object balance skills at 12 weeks.
  YBT requires children to balance on one leg whilst simultaneously reaching as far as possible with the other leg in three separate directions: anterior, posterolateral, and posteromedial. The YBT composite score is calculated by summing the 3 reach directions and normalizing the results to the lower limb length. All measurement scores were taken from scales on standing boards to the nearest 0.5 cm. Distances can be read from the test equipment. Each test was repeated three times, and the maximum range in each direction was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Geok soh, Study Director — Universiti Putra Malaysia
Locations (1):
- Wuyi Road Primary School, Taiyuan City, Shanxi Province, China, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baron J, Bieniec A, Swinarew AS, Gabrys T, Stanula A. Effect of 12-Week Functional Training Intervention on the Speed of Young Footballers. Int J Environ Res Public Health. 2019 Dec 24;17(1):160. doi: 10.3390/ijerph17010160. PMID 31878326
- [Background] James, C. R. (2007). Functional Training for Athletes At All Levels.
- [Background] Boyle, M. (2004). Functional training for sports. Human Kinetics Publishers.
- [Background] Liebenson, C. (2014). Functional training handbook. Lippincott Williams & Wilkins.
- [Result] Heggond, M. S., Suresh, M. M., & Sundar, K. (2020). Impact of functional training on selected motor fitness components of sprinters. Journal of Xi'an University of Architecture & Technology, 12, 649-654.
- [Result] Kovac D, Krkeljas Z, Venter R. Effect of six-week traditional resistance and functional training on functional performance in female netball players. BMC Sports Sci Med Rehabil. 2022 Jan 15;14(1):10. doi: 10.1186/s13102-022-00402-8. PMID 35033152
- [Result] Radcliffe, J. C. (2007). Functional training for athletes at all levels: workouts for agility, speed and power. Simon and Schuster.